CLINICAL TRIAL: NCT06672419
Title: Effectiveness of Tele-Rehabilitation for Fibromyalgia Using AI-Guided Exercise and Computer Vision Combined With Pain Neuroscience Education (FIBRO IA): A Randomized Controlled Trial
Brief Title: Effectiveness of AI-Guided Exercise and Pain Neuroscience Education for Fibromyalgia (FIBROIA)
Acronym: FibroIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Neurociencia Del Dolor (Other)
Collaborators: Universidad San Sebastián (Other); Universidad Santiago de Cali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FibroIA; ID: USS_0003_11-07-2 (Other: Universidad San Sebastián)
Record Dates: First submitted 2024-10-18; First posted 2024-11-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia; Fibromyalgia Syndrome
Keywords: Fibromyalgia; Tele-rehabilitation; Artificial Intelligence; Computer Vision; Pain Neuroscience Education; Randomized Controlled Trial
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This study employs a parallel-group randomized controlled trial (RCT) design. Participants will be randomly assigned to one of two groups: the intervention group, which will receive AI-guided exercise and pain neuroscience education through a tele-rehabilitation platform, or the control group, which will receive standard care for fibromyalgia, including pharmacological treatment and general physical activity recommendations. The study will use a 1:1 randomization ratio and will be conducted remotely. Randomization will be performed using a computer-generated allocation sequence to ensure unbiased group assignment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention (exercise), complete participant blinding is not feasible. However, to minimize performance and expectation bias, the control group utilizes a visually identical digital platform interface ('sham' digital experience). Outcomes Assessors and the Principal Investigator will remain strictly blinded to group allocation until database lock. Treating physiotherapists (Care Providers) managing the platform alerts may be unblinded to ensure safety, but they are not involved in outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Guided Tele-rehabilitation (Experimental): Participants in this arm will receive a 12-week tele-rehabilitation program guided by artificial intelligence (AI) and computer vision technology. The program consists of three personalized exercise sessions per week, delivered remotely and adapted in real time to participants' capabilities and progress. In addition, participants will attend weekly educational sessions focused on pain neuroscience to improve their understanding of chronic pain mechanisms and enhance self-management strategies.
  The intervention is delivered through a visually identical digital platform used by all participants. Supervising physiotherapists monitor progress and provide standardized support but remain blinded to treatment allocation, as only the intervention group receives the active content (AI-guided exercise and PNE).
  Interventions: Other: AI-Guided Exercise and Pain Neuroscience Education
- Usual Care for Fibromyalgia (Active Comparator): Participants in this arm will receive standard care for fibromyalgia, which typically includes pharmacological management such as pain relievers (e.g., paracetamol, tramadol), antidepressants (e.g., amitriptyline, duloxetine), and anticonvulsants (e.g., pregabalin, gabapentin). They will also be provided with general recommendations on physical activity and disease self-management, in line with current clinical guidelines. In addition, participants will use the same digital platform with a visually identical interface, receiving standard, non-specific educational materials and general activity guidance (without AI-guided exercise feedback or pain neuroscience education modules)
  Interventions: Other: Usual Care for Fibromyalgia

INTERVENTIONS:
Other: AI-Guided Exercise and Pain Neuroscience Education — This intervention consists of a 12-week tele-rehabilitation program using AI and computer vision technology to guide personalized exercise sessions (three per week). Exercises are adjusted in real time by the AI system, and participants also attend weekly sessions of pain neuroscience education to develop improved pain management strategies. The program is delivered remotely via a digital platform that is visually identical for all participants. Supervising physiotherapists oversee progress and provide standardized support but remain blinded to group allocation.
  Arms: AI-Guided Tele-rehabilitation
Other: Usual Care for Fibromyalgia — Standard care includes pharmacological management (pain relievers, antidepressants, anticonvulsants) and general recommendations on physical activity and disease management.
  Drug: Pain Relievers - e.g., paracetamol, tramadol
  Drug: Antidepressants - e.g., amitriptyline, duloxetine
  Drug: Anticonvulsants - e.g., pregabalin, gabapentin
  Other: General Physical Activity and Disease Education - recommendations consistent with current clinical guidelines
  Arms: Usual Care for Fibromyalgia

SUMMARY:
This randomized controlled trial will evaluate the effectiveness of a 12-week, home-based telerehabilitation program for adults with fibromyalgia (FM) combining AI-guided exercise with Pain Neuroscience Education (PNE). Fifty participants will be randomized (1:1) to the digital intervention or usual care. The primary outcome is change in pain intensity from baseline to post-intervention (week 13 ± 7 days), with secondary outcomes including physical function and health-related quality of life. Outcome assessors, the principal investigator, and the study statistician will be blinded to group allocation until database lock.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of a 12-week tele-rehabilitation program that integrates artificial intelligence (AI)-guided exercise, computer vision, and pain neuroscience education (PNE) for individuals with fibromyalgia (FM). The study seeks to determine whether this technology-driven approach can reduce pain intensity, improve physical function, and enhance quality of life in a population that frequently experiences limited benefit from conventional treatment strategies.

Intervention

Participants in the intervention group will use a tele-rehabilitation platform that applies AI and computer vision to deliver personalized exercise programs. The AI system monitors performance in real time and adapts exercises to individual capacities and progress. In parallel, participants will attend weekly sessions of pain neuroscience education, designed to improve their understanding of pain processing within the nervous system and to promote more effective self-management through cognitive and behavioral strategies.

The control group will receive standard care for fibromyalgia, which typically includes pharmacological management (e.g., analgesics, antidepressants, anticonvulsants) alongside general recommendations for physical activity and self-care. Comparison between the groups will allow assessment of the added value of combining AI-guided tele-rehabilitation with PNE.

Study Design Participants will be randomly assigned (1:1) to intervention or control group. The intervention will last 12 weeks, during which participants in the intervention group will complete three exercise sessions per week and one educational session weekly. All sessions will be conducted remotely through a user-friendly platform accessible via smartphones or computers. Outcome assessments will be conducted at baseline and immediately after completion of the 12-week program.

Masking: Participants and investigators will remain blinded to group allocation. Outcome assessors and the statistician will also remain blinded until database lock

Objectives

The primary objective is to determine whether the AI-guided exercise and PNE program reduces pain intensity and improves physical function compared with standard care. Secondary objectives include evaluating changes in quality of life, psychological well-being, and treatment adherence. Findings will provide evidence on whether technology-enabled rehabilitation can serve as an accessible, effective alternative for fibromyalgia management.

Rationale

Conventional therapies for fibromyalgia, such as pharmacological treatment and standard physical therapy, often provide suboptimal relief. Tele-rehabilitation represents a promising strategy to deliver personalized, supervised exercise at scale, particularly for patients in underserved or remote areas. When combined with pain neuroscience education, this approach addresses both physical and cognitive aspects of pain, with the potential to improve outcomes beyond current standards of care.

This study aligns with broader public health goals to improve access to effective interventions for chronic pain. Its results may inform future clinical guidelines and support the integration of AI-driven tele-rehabilitation into routine practice for fibromyalgia and related chronic pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia according to the American College of Rheumatology criteria (2016).
* Age between 18 and 65 years.
* Access to an internet-connected device (smartphone or computer).
* Ability to participate in a tele-rehabilitation program.

Exclusion Criteria:

* Participation in another clinical trial in the last 3 months.
* Pregnancy or breastfeeding.
* Uncontrolled severe medical conditions that could interfere with the intervention (e.g., cardiac or pulmonary diseases).
* Physical or cognitive impairments that prevent following the exercise program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analog Scale (VAS) | 12 weeks
  Pain intensity will be measured using the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (worst pain imaginable). Participants will rate their pain at baseline and after 12 weeks of intervention. Higher scores indicate a worse outcome (greater pain intensity). The primary outcome focuses on changes in pain intensity from baseline to the end of the 12-week period.

SECONDARY OUTCOMES:
Change in the Impact of Fibromyalgia on Daily Life Measured by the Revised Fibromyalgia Impact Questionnaire (FIQ-R) | 12 weeks
  The impact of fibromyalgia on daily life will be assessed using the Revised Fibromyalgia Impact Questionnaire (FIQ-R), a tool that measures the overall burden of fibromyalgia on patients through three key domains: overall impact on daily life, severity of specific symptoms, and functional ability in daily tasks. The FIQ-R provides a comprehensive score ranging from 0 to 100, where higher scores reflect a worse outcome (indicating a greater negative impact of fibromyalgia on daily life). This secondary outcome measure will evaluate changes in the total FIQ-R score from baseline to the end of a 12-week intervention period.
Lower Limb Strength and Endurance Measured by the 30-Second Sit-to-Stand Test | 12 weeks
  The 30-second sit-to-stand test measures lower limb strength and endurance by counting the number of times a participant can stand up from a seated position and sit back down within 30 seconds. Higher scores indicate a better outcome (greater strength and endurance). This test serves as a reliable indicator of overall physical function and has been validated for remote use (Bowman et al., 2023). The test will be conducted at baseline and after 12 weeks of intervention.
Change in Quality of Life Measured by EQ-5D | 12 weeks
  Quality of life will be assessed using the EQ-5D (EuroQol-5 Dimension), a standardized measure to evaluate health-related quality of life. The EQ-5D examines five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores range from -0.59 to 1, where higher scores indicate a better quality of life. Scores will be compared from baseline to the end of the 12-week intervention.
Change in Psychological Well-being Measured by the Numeric Rating Scale for Anxiety (NRS-A) | 12 weeks
  The NRS-A is a simple, validated tool that allows patients to rate their level of anxiety on a scale of 0 to 10, where 0 indicates 'no anxiety' and 10 represents 'the worst imaginable anxiety.' Anxiety levels will be measured at baseline and after 12 weeks of intervention.
Perceived Barriers to Treatment Adherence Measured by the Treatment Adherence Barriers Questionnaire | 12 weeks
  The Treatment Adherence Barriers Questionnaire identifies perceived barriers that patients face in adhering to treatment recommendations. This measure provides valuable insights into factors affecting adherence and will be evaluated at baseline and after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Morales-Osorio, PhD, Principal Investigator — Universidad San Sebastian
Locations (2):
- Universidad San Sebastián, Concepción, Región del Biobío, Chile
- Universidad Santiago de Cali, Cali, Colombia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request after publication of the main results. Data will be transferred via secure encrypted platforms and shared in compliance with GDPR and HIPAA regulations. Raw platform data (e.g., motion capture logs, video files) will not be shared due to privacy and technical restrictions."
Supporting Information: Study Protocol
Time Frame: Data will be available after publication of the primary results and for a period of 5 years thereafter.
Access Criteria: vailable upon reasonable request from qualified researchers. A data use agreement will be required.

REFERENCES:
- [Result] Suero-Pineda A, Oliva-Pascual-Vaca A, Duran MR, Sanchez-Laulhe PR, Garcia-Frasquet MA, Blanquero J. Effectiveness of a Telerehabilitation Evidence-Based Tablet App for Rehabilitation in Traumatic Bone and Soft Tissue Injuries of the Hand, Wrist, and Fingers. Arch Phys Med Rehabil. 2023 Jun;104(6):932-941. doi: 10.1016/j.apmr.2023.01.016. Epub 2023 Feb 8. PMID 36758713